CLINICAL TRIAL: NCT04665024
Title: The Effect of Preoperative Chest Physiotherapy on Oxygenation and Lung Functions Among Open Heart Surgery Patients
Brief Title: Effect of Preoperative Chest Physiotherapy on Lung Functions Among Open Heart Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4114.316-474/kk15/2011
Record Dates: First submitted 2020-12-09; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Open Heart Surgery Patients
Keywords: Open heart surgery, chest physiotherapy, spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): G1 included patients undergoing planned surgery who performed chest physiotherapy at home in two weeks period before the surgical operation pre and postoperative chest physiotherapy was performed in G1.
  The chest physiotherapy included the following steps
  1. Snipping through the nose several times, then breathe out through the mouth
  2. Taking a deep breath through the nose, hold the air in, push it down in the stomach, than back to the chest, and in the end breath out through the mouth
  3. Put both hands on the shoulders. Lift the elbows to the sides and take a deep breath through the nose, then lower them, breathe out through the mouth. This procedure was done for the other side as well.
  4. Put both hands on your hips. Lift your right arm to the side, turn backwards with it and take a deep breath through the nose, then turn back, put your hand back to the hip and breathe out through the mouth.This procedure was done for the other side as well
  Interventions: Procedure: preoperative chest physiotherapy; Procedure: postoperative chest physiotherapy
- Group 2 (Active Comparator): G2 included patients who patients undergoing planned surgery but did not perform preoperative chest physiotherapy at home.only postoperative chest physiotherapy made in G2.
  The patient was seen on the first day after surgery in the intensive care unit and was asked if he had performed breathing exercises at home before surgery and then re-evaluation of both groups with respect to respiratory functions and oxygen saturation values from the first day until the seventh after surgery. Also, a daily chest physical therapy program was introduced in accordance with the hospital's policy until the patient's discharge.
  Postoperative chest physiotherapy made in both two groups was similar to the preoperative chest physiotherapy mentioned above but this was achieved by physiotherapists and made once a day for 10-25 minutes depending on the "lectures" of postoperative days.
  The exercises were repeated 10 times and performed 3-4 times per day.
  Interventions: Procedure: postoperative chest physiotherapy

INTERVENTIONS:
Procedure: preoperative chest physiotherapy — The patients were approached to partake in the investigation after they got full clarifications about the point of study. They were allocated into two groups and reassurance was achieved about the absence of any side effects.Furthermore, the examination was approved by the ethical committee.
  Effects of preoperative chest physiotherapy were compared between two groups, by measuring the lung functions, oxygen saturation, pulmonary complications and length of hospital staying. Lung functions were completed by utilizing spirometry parameters, oxygen saturation was measured by pulse oximeter and pulmonary complications were diagnosed by specialist doctors.
  Arms: Group 1
Procedure: postoperative chest physiotherapy — Postoperative chest physiotherapy made in both two groups was similar to the preoperative chest physiotherapy but this was achieved by physiotherapists and made once a day for 10-25 minutes depending on the "lectures" of postoperative days.

SUMMARY:
Postoperative respiratory complications in patients who had chest-opening heart surgery are considered one of the serious factors threatening their life. However, these potential complications could be minimized using proper preoperative chest physiotherapy. This study was designed to assess the potential effects of using preoperative chest physiotherapy on oxygenation and lung functions among open heart surgery patients during postoperative period.

DETAILED DESCRIPTION:
The research was lasted four months in outpatient clinic, cardiothoracic surgical department and intensive care unit at University of Pécs, Clinical Centre, Heart Institute, Hungary . A convenient sample of 100 patients were divided into two groups: group 1 and 2. Group 1 (G1) included patients undergoing planned surgery who performed chest physiotherapy at home in two weeks period before the surgical operation, and group 2 (G2) included patients who patients undergoing planned surgery but did not perform preoperative chest physiotherapy at home. Preoperative and postoperative chest physiotherapy was performed in G1, and only postoperative one made in G2. Potential effects of preoperative chest physiotherapy were studied in both groups with respect to oxygen saturation, pulmonary complications and length of hospital staying. O2 saturation,O2 supplementation, forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) were all measured in a day before (zero day) surgery as well as the first seven days of postoperative period.

Results: Measures of oxygen level and lung functions were significantly (P<0.05) changed in studied groups. The mean values of O2 saturation and supplementation measured in almost seven days of postoperative period were significantly (p<0.05) higher among G1 compared to the values of G2. The same trend was also correct for the mean values of FVC and FEV1.

Conclusions: The results concluded that, the performance of preoperative chest physiotherapy before open heart surgery is recommended, as it might result in the decrease of complications of heart surgery, improvement of respiratory functions and length of staying at hospital.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Under 18 years old; (2) a history of musculoskeletal disorders; (3) patients who had suffered strokes; (4) and psychological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in oxygen saturation | in a day before (zero day) surgery as well as the first seven days of postoperative period.
  Sao2
Change in pulmonary functions | At the first seven days of postoperative period
  FVC and FEV1

SECONDARY OUTCOMES:
pulmonary complications | At the first seven days of postoperative period.
  pneumonia, atelectasis, phrenic nerve stimulation, ventilator
length of hospital staying | The minimum stay for the patient is 7 days
  How many days did the patient stay in the hospital?

CONTACTS AND LOCATIONS:
Overall Officials: VERZAR 7- ZSOFIA, Doctor, Study Director — University of Pecs
Locations (1):
- Heart Institute,Medical School, University of Pécs, Pécs, Pecs, Hungary

REFERENCES:
- [Derived] Shahood H, Pakai A, Rudolf K, Bory E, Szilagyi N, Sandor A, Zsofia V. The effect of preoperative chest physiotherapy on oxygenation and lung function in cardiac surgery patients: a randomized controlled study. Ann Saudi Med. 2022 Jan-Feb;42(1):8-16. doi: 10.5144/0256-4947.2022.8. Epub 2022 Feb 3. PMID 35112592